CLINICAL TRIAL: NCT01213745
Title: A Prospective Randomised Controlled Study to Investigate the Effectiveness of Using a Quality of Life Questionnaire to Target Interventions to Improve Quality of Life in Patients With Lung Cancer
Brief Title: The Use of a Quality of Life Questionnaire in Patients With Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Dr Mary O'Brien, Royal Marsden NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CCR3454
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-10

CONDITIONS: Lung Cancer
Keywords: lung; cancer; quality of life
MeSH Terms: conditions — Lung Neoplasms; Neoplasms | interventions — Methods; Neuropsychological Tests

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention (Experimental)
  Interventions: Other: Intervention
- Attention (Experimental)
  Interventions: Other: Attention
- Control (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention
  Arms: Intervention
Other: Attention
  Arms: Attention
Other: Control
  Arms: Control

SUMMARY:
This study will investigate the effectiveness of using the European Organisation for Research and Treatment of cancer Core Quality of Life Questionnaire (EORTC QLQ-C30 + LC 13) to identify and target therapies in patients with lung cancer. The study will assess whether using the questionnaire will result in an improvement in QoL.

DETAILED DESCRIPTION:
Patients with lung cancer who have completed a course of treatment (or who are in-between treatment) at the Royal Marsden Hospital would be eligible for inclusion in the study. Participants will be randomised into 3 groups. Group 1 - this group will complete the QoL questionnaire and will receive targeted therapies by a doctor (and other members of the oncology team) during a clinic consultation. Group 2 - will complete the QoL questionnaire however the questionnaire will not be seen by the doctor during a clinic consultation. Group 3 - the control group will not complete the QoL questionnaire before a clinic consultation. All patients will complete a diary of all contact they have with health care professionals during the study. The study will last for 6 weeks and at the end of the study all patients will complete the QoL questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* male or female age > 18 years
* patients who are able to adequately understand written and spoken english
* diagnosis of lung cancer (non small cell, small cell, mesothelioma)
* no plan to commence treatment (chemotheraphy, targeted therapies, radioterhapy, surgery) with 6 weeks
* both radically or palliatively treated patients remain eligible
* patients whose toxicities from their primary treatment has resolved or have stabilised for a period of 7 days

Exclusion Criteria:

* patients are taking part on any other QoL studies
* taking part in any other studies that requires QoL questionnaires, extra visits or investigations
* currently on treatment (chemotherapy, radiotherapy, surgery or targeted therapies)
* they have on going toxicities from their treatment which have not been stablised (required intervention within last 7 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
To investigate whether the use of QOL questionnaires during the assessment and management of lung cancer patients results in improved quality of life

SECONDARY OUTCOMES:
To investigate whether the use of EORTC QLQ-C30 + lung cancer module results in less patient contact with health care professionals during the 6 week study period for the 3 groups

CONTACTS AND LOCATIONS:
Overall Officials: Dr M O'Brien, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, United Kingdom

REFERENCES:
- [Derived] Nimako K, Ayite B, Priest K, Severn J, Fries HM, Gunapala R, Bhosle J, Popat S, O'Brien M. A randomised assessment of the use of a quality of life questionnaire with or without intervention in patients attending a thoracic cancer clinic. Eur J Cancer Care (Engl). 2017 Jul;26(4). doi: 10.1111/ecc.12402. Epub 2015 Nov 10. PMID 26556778